CLINICAL TRIAL: NCT05234385
Title: Functional Outcome Following Surgical Treatment of Patients With Sternoclavicular Joint Infection
Acronym: SCJ Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02343; kt22Lardinois
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Sternoclavicular Joint Infection
Keywords: QuickDASH questionnaire; extended SCJ resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Sternoclavicular joints (SCJ) represents an important factor in stability of shoulder joint. Its influence and its function is important for the functionality of the shoulder. SCJ infection is a rare condition and remains often mistreated and potentially life threatening.

This study is to assess the cases treated at the University Hospital Basel with a surgical approach of extended resection of the SCJ. One prospective follow-up visit inclusive one physical examination per patient will be performed to evaluate the long-term functional results of arm, shoulder, hand function with the QuickDASH questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient assigned and treated at the Department of Thoracic Surgery, University Hospital Basel (USB)
* At hospital admission diagnosed with clinical characteristics of sternoclavicular joint infection
* Surgical treatment of extended SCJ resection received
* Signed written informed consent according to ICH-GCP regulations prior to initiation of any protocol-specific activities/procedure
* Patients who died will be included if a signed USB general research consent is available

Exclusion Criteria:

* Isolated sternal or clavicular infection
* Patients received other surgery than extended SCJ resection at USB thoracic surgery
* Inability to follow procedures or insufficient knowledge of language (German/French) or inability to give consent
* Patients who have clearly stated that they would not agree in providing their clinical data for scientific purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with SCJ infection and surgical treatment of extended SCJ resection, treated at the Department of Thoracic Surgery at the University Hospital Basel between 31.05.2011 and 28.02.2022.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
QuickDASH score | one time assessment at the prospective follow-up visit (timeframe of maximal 1 hour)
  QuickDASH score of the mobility of the arm, shoulder, hand and its function by using the QuickDASH questionnaire. The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (4 items, scored 1-5). A higher score indicates greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. Dr. med., Study Director — Department of Thoracic Surgery, University Hospital Basel
Locations (1):
- Department of Thoracic Surgery, University Hospital of Basel, Basel, Switzerland

REFERENCES:
- [Result] Vujic J, Hojski A, Dackam SVC, Bachmann H, Lardinois D. Functional Outcomes of Patients With Sternoclavicular Joint Infection After Extended Resection. Ann Thorac Surg Short Rep. 2024 Jan 19;2(2):193-196. doi: 10.1016/j.atssr.2023.12.015. eCollection 2024 Jun. PMID 39790151